CLINICAL TRIAL: NCT06921122
Title: Use Of The Iowa Oral Performance Instrument In Speech Therapy Intervention In Individuals With Parkinson's Disease: Randomized Clinical Trial
Brief Title: Use Of A Tongue Strength Training Device And Its Relationship With Speech In Patients With Parkinson's Disease
Acronym: IOPI
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Collaborators: Federal University of Rio Grande do Sul (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20240194
Record Dates: First submitted 2025-03-06; First posted 2025-04-10 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Parkinson Disease (PD)
Keywords: Dysarhria; Speech Therapy; IOPI; Intervention; Parkinson Disease (PD)
MeSH Terms: conditions — Parkinson Disease; Communication Disorders | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Iopi (Experimental): All individuals will perform a program of two lingual exercises: the first exercise consists of compressing the air-filled bulb between the tongue and the anterior portion of the hard palate using IOPI, in order to sustain the articulatory positioning for "p" (closed lips) and "t" (tongue tip behind upper teeth) and hold for 4 seconds. The second exercise consists of compressing this same bulb between the tongue and the posterior portion of the hard palate, performing 10 repetitions, 3 times a day on 3 days of the week, as recommended for strength training by the American College of Sports Medicine. These tongue locations were selected based on evidence of regional differences in lingual muscle composition, marked by a higher percentage of muscle tissue in the posterior region of the tongue that may respond differently to exercise.
  Interventions: Device: IOWA ORAL PERFORMANCE INSTRUMENT
- Placebo (Placebo Comparator): The study group, without treatment, evaluated on the same schedule as treated patients, will represent the natural progression of speech disorders in PD. The decision was made not to include a sham treatment, in order to adhere to the principle of balance and not place an undue burden of time and effort on patients who received a treatment with low therapeutic potential. Furthermore, the investigators considered that given questions about the suitability of simulations as treatment comparators in behavioral studies, the research in this work between study group and placebo group (no treatment) may provide more useful contrasts than a therapeutic simulation group.
  If an intervention proposal is proven to bring direct benefits to the participants, this group will be contacted to carry out the same intervention later.
  Interventions: Device: Placebo Group - Without Treatment

INTERVENTIONS:
Device: IOWA ORAL PERFORMANCE INSTRUMENT — In the first session all protocols and assessments will be carried out as a way of observing the responses and previous measures of all participants. The group in this study must appear weekly for six weeks to verify if necessary, reinsufflate the bulb, carry out force measurement and lingual press with the IOPI, as well as receive or reinforce the guidance provided at the beginning of the treatment.
  The participants in the group will study that will have a mobile phone and an instant message application will receive weekly, on scheduled days, a letter containing the following text message: "Here is the day of performing the last exercise by the Speech Pathologist". Participants who do not have a mobile phone will be notified through a telephone connection or contact with a responsible family member/caregiver.
  After the end of the sixth week of training, patients will be subjected to the last set of data on the two protocols and evaluations proposed in this study.
  Arms: Iopi
Device: Placebo Group - Without Treatment — The group in study, without treatment, supported by the same schedule of the patients treated, will represent the natural progression of failure disorders in PD. A decision was made not to include a false treatment, in order to adhere to the principle of balance and not to place an undue burden of time and effort on patients who receive a treatment with low therapeutic potential. Furthermore, the researchers considered that given the questions regarding the adequacy of simulations as comparators of treatment in behavioral studies, research in this work between the group in the study and the placebo group (without treatment) can provide more useful contrasts than a group with therapeutic simulation.
  If the intervention clearly aims to provide direct benefits to the participants, this group will be contacted to carry out the same intervention later.
  Arms: Placebo

SUMMARY:
Parkinson's Disease affects the brain and causes several movement problems. These problems include stiff muscles, slow movements, shaking when resting, and trouble keeping balance. As the disease gets worse, it can also affect how people speak.

Doctors and therapists have found better ways to test how Parkinson's affects speech. There's one special therapy method that's considered the best for helping people with Parkinson's speak better. Now, they're also using a new tool called IOPI (Iowa Oral Performance Instrument) to help test and treat speech problems.

This research project wants to see if using IOPI can help people with Parkinson's speak better. Here's how they'll do it:

First, they'll split people with Parkinson's into two groups randomly. Everyone will take speech tests, like:

Holding an "a" sound as long as they can; Saying "pataka" repeatedly; Counting from 1 to 15; Reading sentences; Speaking freely about a topic; They'll also measure how strong their tongue is using IOPI. Then, one group will get therapy using the IOPI tool, while the other group won't. After the therapy is done, they'll test everyone again to see if the IOPI therapy helped improve their speech.

The researchers hope this study will show that IOPI is a helpful new tool for speech therapy, giving therapists more ways to help people with Parkinson's speak better.

DETAILED DESCRIPTION:
Characterized by dopaminergic neurodegeneration, Parkinson's Disease (PD) manifests various motor symptoms, including: rigidity, bradykinesia, resting tremor, and postural instability, which impact the speech of affected individuals as they progress. Considerable advances have been made regarding speech assessment methods, and a globally recognized intervention model is used as the gold standard for speech-language therapy in individuals with Parkinson's Disease. However, currently, instruments such as the IOPI (Iowa Oral Performance Instrument Measures) have been gaining ground in the assessment and therapy of these subjects. Thus, this work aims to apply an intervention model for speech therapy in PD patients using IOPI as a treatment tool through a randomized clinical trial. This study will consist of three phases: The first phase will consist of random allocation of subjects between control and intervention groups. Sequentially, all subjects will undergo speech assessment using speech tasks: maximum phonation time through sustained vowel /a/, diadochokinesis of alternating syllables /pataka/, counting numbers from 1 to 15, sentence reading, and monologue, then IOPI will be used to verify the tongue pressure of participating subjects. The second phase will encompass therapy with the IOPI instrument in the intervention group, and the third phase will be the reassessment of subjects from both groups. It is considered that the findings of this study may contribute to the addition of new instruments to therapy and, thus, provide new approaches and expansion of the therapeutic perspective for the speech of subjects with PD.

ELIGIBILITY:
Inclusion Criteria:

* All individuals with an age greater than or equal to 18 years who have been diagnosed with idiopathic PD attended at the Movement Disorders Outpatient and at the Speech Therapy Outpatient Degenerative Adult of a quaternary health care hospital.
* Who will participate in the project entitled Validation and applicability of the Test of Mastication and Swallowing Solids (TOMASS) for the Brazilian population with Parkinson's disease approved under No. 2023-0402.

Exclusion Criteria:

* Subjects who are not currently off the medication;
* Those whose serious alterations of language and cognition are unable to perform the proposed tasks;
* Those with other neurological conditions will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-04-10 (Estimated); Primary Completion 2026-12-20 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
Effect of IOPI on the articulatory subsystem | 6 weeks
  The investigator determines the safe target value for therapy purposes and provides specific instructions to the subject. The target value definition will be expressed by means of an algebraic formula, based on the internationally recognized unit of pressure, the Pascal (Pa).
  Strength is measured with the IOPI by quantifying the length of time that a patient can maintain 50% of his or her maximum pressure. This procedure is conducted by setting the target value in the Target Mode to 50% of the patient's maximum pressure and timing how long the patient can hold the top (green) light on.
  There is considerable variability in tongue strength in a population of adults reporting no swallowing or speech problems. There is a clear central tendency, however, with an average maximum pressure of about 60 kPa, and a range of 40-80 kPa.

SECONDARY OUTCOMES:
Sociodemographic Variables | 6 weeks
  The secondary objectives include correlating speech articulation data and IOPI training with variables such as age, sex, disease duration, and age at symptom onset. These variables will be collected through the application of a sociodemographic questionnaire. If the findings demonstrate a positive correlation, this may indicate the need for early speech therapy intervention in these patients, preventing the necessity of waiting for the disease to progress to more advanced stages.

OTHER OUTCOMES:
Unified Parkinson's Disease Rating Scale III - UPDRS III | 6 weeks
  The Unified Parkinson's Disease Rating Scale is composed of four parts, which assess different aspects of PD manifestations. Items receive values between 0 (normal) and 4 (severe). Part III - motor assessment - was chosen for the purposes of this study and the score will be collected by checking data from the electronic medical record.
Radboud Oral Motor Inventory for Parkinson's Disease - ROMP | 6 weeks
  ROMP is a self-assessment protocol for three domains: speech, swallowing and saliva. It consists of 23 items, seven items corresponding to the speech domain, seven items for swallowing and nine items related to saliva. The patient marks the frequency of symptoms from 1 to 5 (1 = normal; 5 = worst score). The minimum total score is 23 and the maximum score is 115 points. In this work, only the self-assessment of the speech domain will be applied, to determine whether patients can perceive changes in their speech, even subtle ones.

CONTACTS AND LOCATIONS:
Overall Officials: Amanda L Bressanelli, Academic, Study Director — Federal University of Rio Grande do Sul; Vitória M Santos, Academic, Study Chair — Federal University of Rio Grande do Sul; Maira R Olchik, Teacher, Principal Investigator — Federal University of Rio Grande do Sul
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Product Description — https://iopimedical.com/